CLINICAL TRIAL: NCT04690751
Title: Relative Bioavailability of a Single 200 MG Dose Of Cenobamate (YKP3089) Given As An Oral Tablet Or As An Oral Suspension And The Effect Of Food On A Single 200 MG Dose Of Cenobamate Given As An Oral Suspension
Brief Title: Bioavailability and Food Effect Study of Cenobamate as an Oral Suspension and Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YKP3089C037
Record Dates: First submitted 2020-12-10; First posted 2020-12-31 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — Cenobamate

STUDY DESIGN:
Intervention Model Description: • This study is an open-label, randomized, single-dose, single-center, three-period, six-sequence, balanced crossover study in healthy male and female subjects to assess the relative bioavailability of 200 mg of cenobamate given as an oral tablet or oral suspension and to evaluate the effect of food on the bioavailability of a 200 mg dose of cenobamate given as an oral suspension in fasting and fed conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): Treatment A: Oral Dose of cenobamate administered as a single 200 mg tablet under fasted conditions
  Interventions: Drug: Cenobamate 200Mg Tab Fasted
- Treatment B (Experimental): Treatment B: Oral Dose of cenobamate administered as a single 200 mg/20 mL suspension under fasted conditions
  Interventions: Drug: Cenobomate Oral Suspension Fasted
- Treatment C (Experimental): Treatment C: Oral Dose of cenobamate administered at a single 200 mg/20 mL suspension under fed conditions
  Interventions: Drug: Cenobamate Oral Suspension Fed

INTERVENTIONS:
Drug: Cenobamate 200Mg Tab Fasted — Cenobamate (YKP3089) is a small molecule approved in the United States (US) for the treatment of partial onset seizures (POS) in adult patients.
  Other Names: YKP3089
  Arms: Treatment A
Drug: Cenobamate Oral Suspension Fed — Cenobamate (YKP3089) is a small molecule approved in the United States (US) for the treatment of partial onset seizures (POS) in adult patients.
  Other Names: YKP3089
  Arms: Treatment C
Drug: Cenobomate Oral Suspension Fasted — Cenobamate (YKP3089) is a small molecule approved in the United States (US) for the treatment of partial onset seizures (POS) in adult patients.
  Other Names: YKP3089
  Arms: Treatment B

SUMMARY:
This study is designed to evaluate the relative bioavailability, or the degree and rate at which the drug is absorbed by the body of two cenobamate formulations (200 mg Oral Suspension and a 200 mg Oral Tablet) and to assess the effect of food on the oral bioavailability of the 200 mg Oral Suspension. This study will also look at the safety and tolerability of the oral suspension and the oral tablet under both fasted and fed conditions.

DETAILED DESCRIPTION:
This study is an open-label, randomized, single-dose, single-center, three-period, six-sequence, balanced crossover study in healthy male and female subjects to assess the relative bioavailability of 200 mg of cenobamate given as an oral tablet or oral suspension and to evaluate the effect of food on the bioavailability of a 200 mg dose of cenobamate given as an oral suspension in fasting and fed conditions.

The study consists of a 28-day screening period, followed by single dose administration of cenobamate (tablet or suspension) on Day 1, Day 22, and Day 43, an assessment period of 62 days and a follow-up visit on Day 69. All subjects will be confined to the clinical site from Day -1 (the day before period 1 dosing) until the morning of Day 4, Day 20 (the day of the last PK sampling for period 1) until the morning of Day 25, and Day 41 (the day of the last PK sampling for period 2) until the morning of Day 46. Outpatient visits will be performed regularly until the 456-hour PK sampling for each period. The follow-up visit will occur on Day 69 (±1 day).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects of 18 to 50 years of age (inclusive), at the time of screening
2. Able to read, understand, sign, and date a written informed consent form (ICF) before study participation at screening
3. Agree to use effective methods of contraception as described in Section 12.1.7.8 and Section 12.1.7.9.
4. Body mass index (BMI) between 18.5 and 30.0 kg/m2 (inclusive) at screening
5. Judged to be in good health on the basis of medical history, physical examination, and routine laboratory measurements (i.e., without clinically relevant pathology)
6. Electrocardiogram (ECG) (12-lead), arterial blood pressure, and heart rate within the normal range of the study center or considered not clinically significant by the Investigator.
7. Able to understand and comply with protocol requirements and instructions and likely to complete the study as planned
8. Females of non-childbearing potential (18 to 50 years of age (inclusive)), who have undergone a sterilization procedure at least 6 months prior to dosing with official documentation (e.g., bilateral tubal ligation or bilateral salpingectomy or hysterectomy), or be postmenopausal with amenorrhea for at least 1 year prior to dosing and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status as per Principal Investigator's judgment

Exclusion Criteria:

1. Clinically relevant abnormal medical history, abnormal findings on physical examination, vital signs, ECG, or laboratory tests at Screening that the Investigator judges as likely to interfere with the objectives of the trial or the safety of the volunteer
2. Smokers (subjects who have smoked within 6 months at screening)
3. History of any drug related hypersensitivity reactions as well as severe hypersensitivity reactions (like angioedema) or DRESS as evaluated by the Investigator
4. Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with pharmacokinetics of the study drug (except appendectomy and simple hernia repair)
5. Any prescribed or over-the-counter medication taken within 2 weeks prior to start of administration of study drug (Day 1) or within 6 times the elimination half-life of the medication prior to start of study drug intake (whichever is longer). Occasional use of acetaminophen is allowed up until 24 hours before dosing
6. Consumption of herbal medications, dietary supplements and specific fruit products. Subjects should have stopped consumption of herbal medications or dietary supplements (e.g., St. John's Wort, ginkgo biloba, and garlic supplements), and grapefruit or grapefruit juice, or Seville oranges at least 2 weeks before the first dosing day of study drug. Vitamins/mineral supplements are allowed up until 24 hours before dosing
7. History of drug or alcohol abuse or addiction within 2 years before the start of study drug dosing, or a positive test results for alcohol or drugs of abuse, such as amphetamine, barbiturate, benzodiazepine, cocaine, methadone, opiates, oxycodone, phencyclidine, propoxyphene, cannabinoid (THC), MDMA (Ecstasy), methaqualone, and tricyclic antidepressant (TCA)
8. Regular consumption of more than 2 units of alcoholic beverages per day or more than 14 units per week (1 unit of alcohol equals 1 pint [473 mL] of beer or lager, 1 glass [125 mL] of wine, 25 mL shot of 40% spirit) before screening
9. Consumption of an average of more than 5 servings (8 ounces per serving) per day of coffee, cola, or other caffeinated or methyl xanthine beverages before screening
10. Consumption of any caffeine- or methyl xanthine-containing products (e.g., coffee, tea, chocolate, or soda) or alcoholic beverages within 48 hours prior to Day 1 of each period and until the end of each PK sampling period
11. Participation in a clinical study involving administration of either an investigational or a marketed drug within 2 months or 7 half-lives (whichever is longer) before screening
12. Blood donation or a significant loss of blood within 60 days of the start of study drug dosing or donation of more than 1 unit of plasma within 7 days before screening
13. Positive result at screening for any of the following infectious disease tests: hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), human immunodeficiency virus antigen and antibody (HIV Ag, HIV Ab)
14. Illness within 5 days before the start of study drug dosing ("illness" is defined as an acute [serious or non-serious] condition [e.g., the flu or the common cold])
15. History of any known relevant allergy/hypersensitivity (including allergy to the trial medication or its excipients)
16. Subject who is judged not eligible for study participation by Investigator
17. History of Familial Short QT syndrome.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Greene, PharmD, Study Chair — SK Life Science, Inc.
Locations (1):
- PRA Health Sciences Salt Lake City, Millcreek, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Treatment ABC, with 21 day washout periods between each dose. Treatment A: Oral Dose of cenobamate administered as a single 200 mg tablet under fasted conditions Treatment B: Oral Dose of cenobamate administered as a single 200 mg/20 mL suspension under fasted conditions Treatment C: Oral Dose of cenobamate administered at a single 200 mg/20 mL suspension under fed conditions
- Sequence 2: Treatment BCA, with 21 day washout periods between each dose. Treatment A: Oral Dose of cenobamate administered as a single 200 mg tablet under fasted conditions Treatment B: Oral Dose of cenobamate administered as a single 200 mg/20 mL suspension under fasted conditions Treatment C: Oral Dose of cenobamate administered at a single 200 mg/20 mL suspension under fed conditions
- Sequence 3: Treatment CAB, with 21 day washout periods between each dose. Treatment A: Oral Dose of cenobamate administered as a single 200 mg tablet under fasted conditions Treatment B: Oral Dose of cenobamate administered as a single 200 mg/20 mL suspension under fasted conditions Treatment C: Oral Dose of cenobamate administered at a single 200 mg/20 mL suspension under fed conditions
- Sequence 4: Treatment ACB, with 21 day washout periods between each dose. Treatment A: Oral Dose of cenobamate administered as a single 200 mg tablet under fasted conditions Treatment B: Oral Dose of cenobamate administered as a single 200 mg/20 mL suspension under fasted conditions Treatment C: Oral Dose of cenobamate administered at a single 200 mg/20 mL suspension under fed conditions
- Sequence 5: Treatment BAC, with 21 day washout periods between each dose. Treatment A: Oral Dose of cenobamate administered as a single 200 mg tablet under fasted conditions Treatment B: Oral Dose of cenobamate administered as a single 200 mg/20 mL suspension under fasted conditions Treatment C: Oral Dose of cenobamate administered at a single 200 mg/20 mL suspension under fed conditions
- Sequence 6: Treatment CBA, with 21 day washout periods between each dose. Treatment A: Oral Dose of cenobamate administered as a single 200 mg tablet under fasted conditions Treatment B: Oral Dose of cenobamate administered as a single 200 mg/20 mL suspension under fasted conditions Treatment C: Oral Dose of cenobamate administered at a single 200 mg/20 mL suspension under fed conditions
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 4 | 5 | 5 | 4 | 6 | 4
Completed | 4 | 4 | 4 | 3 | 3 | 4
Not Completed | 0 | 1 | 1 | 1 | 3 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Positive urine drug screen test | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence 1: Treatment ABC, with 21 day washout periods between each dose.
  Treatment A: cenobamate 200 mg oral tablet fasted Treatment B: cenobamate 200 mg/20 mL oral suspension fasted Treatment C: cenobamate 200 mg/20 mL oral suspension fed
- Sequence 2: Treatment BCA, with 21 day washout periods between each dose.
  Treatment A: cenobamate 200 mg oral tablet fasted Treatment B: cenobamate 200 mg/20 mL oral suspension fasted Treatment C: cenobamate 200 mg/20 mL oral suspension fed
- Sequence 3: Treatment CAB, with 21 day washout periods between each dose.
  Treatment A: cenobamate 200 mg oral tablet fasted Treatment B: cenobamate 200 mg/20 mL oral suspension fasted Treatment C: cenobamate 200 mg/20 mL oral suspension fed
- Sequence 4: Treatment CBA, with 21 day washout periods between each dose.
  Treatment A: cenobamate 200 mg oral tablet fasted Treatment B: cenobamate 200 mg/20 mL oral suspension fasted Treatment C: cenobamate 200 mg/20 mL oral suspension fed
- Sequence 5: Treatment ACB, with 21 day washout periods between each dose.
  Treatment A: cenobamate 200 mg oral tablet fasted Treatment B: cenobamate 200 mg/20 mL oral suspension fasted Treatment C: cenobamate 200 mg/20 mL oral suspension fed
- Sequence 6: Treatment BAC, with 21 day washout periods between each dose.
  Treatment A: cenobamate 200 mg oral tablet fasted Treatment B: cenobamate 200 mg/20 mL oral suspension fasted Treatment C: cenobamate 200 mg/20 mL oral suspension fed
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Total
Number analyzed (Participants) | 4 | 5 | 5 | 4 | 6 | 4 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (4.32) | 35.6 (11.67) | 30.6 (12.92) | 29.5 (8.74) | 28.5 (8.17) | 31.0 (5.48) | 30.6 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 0 | 1 | 1 | 5
  Male | 3 | 4 | 4 | 4 | 5 | 3 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 1 | 1 | 2 | 7
  Not Hispanic or Latino | 3 | 3 | 5 | 3 | 5 | 2 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 0 | 0 | 2
  White | 4 | 2 | 5 | 3 | 6 | 3 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 5 | 4 | 6 | 4 | 28
Weight [Mean (Standard Deviation); unit: kg] | 74.45 (6.982) | 73.30 (10.458) | 77.52 (9.785) | 83.38 (10.779) | 72.93 (13.896) | 77.93 (13.178) | 76.24 (10.795)
Height [Mean (Standard Deviation); unit: cm] | 174.93 (9.016) | 173.36 (8.993) | 180.72 (5.404) | 182.00 (0.469) | 172.13 (11.965) | 174.60 (13.879) | 176.05 (9.371)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 24.30 (1.128) | 24.38 (3.047) | 23.76 (2.919) | 25.15 (3.360) | 24.47 (3.133) | 25.58 (3.336) | 24.56 (2.726)

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Maximum observed plasma concentration of cenobamate
Time Frame: 120, 192, 264, 360, 456, hours post-dose
Measure: Median (Full Range); unit: (μg/mL)
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 25 | 24 | 25
(μg/mL) | 4.880 [3.77 to 6.66] | 4.680 [3.81 to 6.56] | 3.860 [3.25 to 4.75]

2. Primary Outcome: Tmax
Description: Time to reach Maximum observed plasma concentration of cenobamate
Time Frame: 120, 192, 264, 360, 456 hour post-dose
Measure: Median (Full Range); unit: (h)
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 25 | 24 | 25
(h) | 3.000 [0.50 to 5.00] | 0.750 [0.50 to 3.50] | 5.000 [3.00 to 10.00]

3. Primary Outcome: Area Under the Concentration Curve to Last Measurable Concentration
Description: AUC from the time of dosing to the time of the last measurable concentration of cenobamate
Time Frame: 120, 192, 264, 360, 456 hour post-dose
Measure: Median (Full Range); unit: (μg•h/mL)
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 25 | 24 | 25
(μg•h/mL) | 304.0 [178 to 516] | 302.5 [165 to 493] | 277.0 [17 to 494]

4. Primary Outcome: Area Under the Concentration Curve From 0 to Infinity
Description: Area Under the Concentration Curve (AUC) from time 0 extrapolated to infinity
Time Frame: 120, 192, 264, 360, 456 hour post-dose
Measure: Median (Full Range); unit: (μg•h/mL)
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 25 | 24 | 25
(μg•h/mL) | 308.0 [183 to 526] | 309.5 [178 to 500] | 296.0 [178 to 500]

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: To evaluate the safety and tolerability of each cenobamate formulation administered under either fed (Oral Dose of cenobamate administered at a single 200 mg/20 mL suspension ) or fasted (Both tablet and oral suspension formulations) incidence of treatment-emergent adverse events will be monitored.
Time Frame: Day 1 to Day 69
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 25 | 24 | 25
Participants | 8 | 8 | 7

ADVERSE EVENTS:
Time Frame: 69 days
Arm/Group | Treatment A | Treatment B | Treatment C
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 8/25 | 8/24 | 7/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=25) | Treatment B (N=24) | Treatment C (N=25)
Paraesthesia Oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter Site Related Reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Euphoric Mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruitus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pseudofolliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT04690751/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT04690751/SAP_001.pdf